CLINICAL TRIAL: NCT02648295
Title: Effects of IV Tranexamic Acid on the Thromboelastogram in Patients Undergoing Total Hip or Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: West Virginia University (Other)
Responsible Party: Principal Investigator, Matthew Dietz, MD, Assistant Professor, West Virginia University
Other Study IDs: 1509851949
Record Dates: First submitted 2015-12-18; First posted 2016-01-07 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Status Post Total Hip and Knee Arthroplasty

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Effects of IV TXA on TEG in patients undergoing THA or TKA — Subjects will undergo surgery per standard of care. All subjects will have 3 additional vials of blood drawn to evaluate TEG.

SUMMARY:
Blood management is an important part of successful total joint replacement. Loss of blood and transfusion can lead to poor outcomes for patients. The use of tranexamic acid (TXA) has become a standard component to many blood management programs. It is used to treat or prevent excessive blood loss during surgery and in various medical conditions such as excessive bleeding or hemorrhage. A normal body process prevents blood clots that occur naturally from growing and causing problems. When this process becomes overactive it can result in excessive bleeding, leading to increased blood transfusions. The proposed study seeks to evaluate the relationship between TXA and thromboelastogram (TEG) results.

ELIGIBILITY:
Inclusion Criteria:

* Primary total hip and knee arthroplasty patients presenting to WVU Center for Joint Replacement
* 40-90 years old

Exclusion Criteria:

* Known coagulopathy
* History of venothrombotic event
* Unstable angina
* Recent Myocardial infarction (MI)
* History of bleeding events
* History of chronic anemia
* Preoperative anemia
* Current use of blood thinners including aspirin

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults undergoing primary total hip and knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
All time measurements which indicate various aspects of clotting cascade | 3 months
  Data derived from the TEG which includes R, MA, LY30 (R = clotting factors, MA clot strength and platelet function and LY30 is fibrinolysis).

SECONDARY OUTCOMES:
Blood loss and transfusions | 3 months
  Estimated and Calculated blood loss and transfusion requirements